CLINICAL TRIAL: NCT06038136
Title: Post-Stroke Enhancement of Delirium Outcomes With Reduction in Neuro-checks
Acronym: SNDOWN
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting grant funding
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00130444
Record Dates: First submitted 2023-08-15; First posted 2023-09-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Delirium; Neuro: Cerebrovascular Accident
MeSH Terms: conditions — Stroke; Ischemic Stroke; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Neuro Checks (No Intervention): If a patient is randomized to the control group, they will continue to have neuro-checks conducted every 2-4 hours as ordered by the primary team, as per standard of care on the acute stroke service.
- Absence of Neuro Checks (Experimental): If a patient is randomized to the intervention group, the team will discontinue neuro-checks between 8pm and 4am. They will otherwise receive the same care, including overnight vital signs. If the patient has a neurologic or hemodynamic change, the primary team may elect to restart the overnight neuro-checks.
  Interventions: Behavioral: Decreased Neuro Checks overnight

INTERVENTIONS:
Behavioral: Decreased Neuro Checks overnight — If a patient is randomized to the intervention group, the team will discontinue neuro-checks between 8pm and 4am. They will otherwise receive the same care, including overnight vital signs. If the patient has a neurologic or hemodynamic change, the primary team may elect to restart the overnight neuro-checks.
  Arms: Absence of Neuro Checks

SUMMARY:
There have been limited studies on delirium in patients hospitalized with acute stroke. There have been no studies on the potential impact of overnight neuro-checks and resulting sleep disruption on delirium or other outcomes. Additional research is needed to determine if overnight checks are necessary or even harmful. We aim to find out if stopping overnight neuro checks may prevent delirium and benefit the patient.

DETAILED DESCRIPTION:
This study hopes to challenge the clinical paradigm that all patients with acute stroke need around-the-clock neuro-checks. The practice of conducting an NIHSS every 4 hours on patients with acute stroke has never been validated, particularly in clinically stable patients, but is the standard of care. This practice potentially comes at the cost of inducing delirium due to poor sleep which can result in numerous adverse outcomes.

This study hopes to identify the impact of eliminating overnight neuro-checks and prioritize sleep and rest. We hypothesize that increased emphasis on sleep will reduce the incidence of delirium and thereby improve the deleterious effects of delirium such as prolonged length of stay and increased likelihood of being discharged to a facility.

A quality improvement project was undertaken to at MUSC to begin to understand the impact of eliminating overnight neuro-checks. This project was focused on patients on the Inpatient Stroke Service, admitted to 9 East. Starting in October 2022, the Stroke team would identify patients who were medically and neurologically stable and place an order to discontinue overnight neuro-checks. Incidence of delirium, LOS, NIHSS, and mRS were compared using data from 4 months prior (June-September 2022) and 8 months after initiation of the project. Compared to pre-intervention, there was a reduction in patients who were delirious from 34-24% and a reduction in average length of stay by 1.5 days. This preliminary data suggests a positive impact of the intervention. There was no change in NIHSS at discharge or the mRS at discharge suggesting there was no negative impact on the patient's neurologic function by eliminating overnight neuro-checks.

The data collect from this preliminary study is exciting, however, warrants more a more scientific evaluation. The proposed study will be a randomized control trial that will help answer these questions more definitively.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with acute stroke Age greater or equal to 18 years old Medical and neurologic stability for discontinuation of neuro-checks, determined by the Stroke Service NP and Attending Physician (no uncontrolled fluctuation in vital signs, seizure like activity or worsening neurologic function) Ability to give informed consent, or identifiable surrogate decision maker

Exclusion Criteria:

Surgical hemorrhagic stroke Subarachnoid hemorrhage Medical or neurologic instability Pregnancy Inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium as measured as change in Confusion Assessment Method (CAM) | From date of randomization until date of hospital discharge, up to 8 weeks
  The Confusion Assessment Method (CAM) is a standardized evidence-based tool that enables non-psychiatrically trained clinicians to identify and recognize delirium quickly and accurately in both clinical and research settings. The CAM includes four features found to have the greatest ability to distinguish delirium from other types of cognitive impairment. A positive or negative result depends on four criteria:
  1. Acute onset and fluctuating course Determined by collateral history or repeated clinic assessment
  2. Inattention Counting from 20-1 is a simple (if blunt) test for this
  3. Disorganised thinking
  4. Altered levels of consciousness The CAM is considered to be positive for the presence of delirium if both features 1 and 2 are present, with at least one of features 3 or 4.The primary outcome will be incidence of delirium as measured as CAM positivity at any point during the hospitalization.

SECONDARY OUTCOMES:
Mean Length of Stay | From date of hospital admission to date of hospital discharge, up to 8 weeks
  Average hospitalization (measured in days)
Change in National Institutes of Health Stroke Scale (NIHSS) Score | From date of hospital admission to date of hospital discharge. From date of hospital discharge to date of 1month follow up appointment. From date of hospital discharge to date of 3 month follow up appointment.
  The scale measures the severity of symptoms associated with patient's stroke. It assesses the severity of impairements related to stroke. The impairments are graded on a 3-4 point scale wtih scores that range from 0-42. Patients with a higher score have a more severe impauirment, and patients with a lower score have a less severe impairment.
Modified Rankin Scale | Within 24 hours of hospital admission, within 24 hours of hospital discharge and at 90 day stroke clinic follow up
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
Discharge Disposition | On date of hospital discharge , up to 8 weeks from randomization
  Location patients are discharged to from the hospital (home vs rehab)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No